CLINICAL TRIAL: NCT03375476
Title: Evaluation of a Model for Post-anesthesia Troponin Increase and Heart Injury Estimation
Acronym: EMPATHIES
Status: Completed | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Tommaso Fossali (Other); Beatrice Borghi (Unknown); Emanuele Catena (Unknown); Andrea Perotti (Unknown)
Responsible Party: Principal Investigator, Riccardo Colombo, Principal Investigator, ASST Fatebenefratelli Sacco
Other Study IDs: PMI_1
Record Dates: First submitted 2017-12-04; First posted 2017-12-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Myocardial Ischemia
Keywords: postoperative myocardial infraction; myocardial injury; general anesthesia; vascular surgery; surgical stress; surgical plethysmographic index
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vascular surgical patients: Patients undergoing elective vascular non-cardiac surgery in general anesthesia
  Interventions: Diagnostic Test: collection of cardiovascular risk scores and intraoperative cardiovascular parameters; Diagnostic Test: cardiac troponin assay; Diagnostic Test: Electrocardiogram

INTERVENTIONS:
Diagnostic Test: collection of cardiovascular risk scores and intraoperative cardiovascular parameters — collection of preoperative cardiovascular risk scores and intraoperative cardiovascular parameters
Diagnostic Test: cardiac troponin assay — plasmatic concentration of high sensitive cardiac troponin will be measured at baseline and on postoperative day 1, 2 and 3
Diagnostic Test: Electrocardiogram — 12 derivations ECG will be made at baseline and on postoperative day 1, 2, and 3

SUMMARY:
This study evaluates the preoperative cardiovascular risk, the intraoperative hemodynamic characteristics and the surgical photo-plethysmographic index of patients undergoing general anesthesia for non-cardiac vascular surgery to develop a multiple variable model assessing the risk for postoperative myocardial ischemic events.

DETAILED DESCRIPTION:
Perioperative cardiac troponin leak is common and is strongly associated with mortality even in absence of classic myocardial infarction signs. In the VISION study 11.6% of patients undergoing non-cardiac surgery were troponin positive and 1.9% (95%CI 1.7-2.1%) of those patients died within 30 days of surgery. In selected populations of patients undergoing vascular surgery, a postoperative cTn leak, without clinical features of myocardial ischemia, is associated with an increased risk of 30-day mortality (odds ratio 5.03, 95% CI 2.88-8.79). Myocardial oxygen supply-demand imbalance and plaque rupture/thrombosis are the main mechanism involved in the pathogenesis of postoperative myocardial ischemic events. Frequently cardiac troponin leaks occur in absence of classical signs and symptoms of myocardial infarction. More than 80% of patients with postoperative cardiac troponin leak are clinically asymptomatic for myocardial ischemia, and ischemic ECG changes are often absent.

The identification of patients who will experience a postoperative myocardial ischemia will continue to be a challenge for anaesthesiologists.The current tool used for risk stratification using the AHA/ACC algorithm is Lee's Revised Cardiac Risk Index. Unfortunately, this tool can only reliably exclude low-risk patients and cannot identify patients which are likely to have perioperative cardiovascular complications.

The surgical plethysmographic index (SPI, GE Healthcare, Finland) during general anaesthesia has been correlated with the stressors of surgery (e.g. intubation, incision, …), and with stress hormone production. It has been demonstrated that SPI and other pulse photo-plethysmographic indices reflect sympathetic-mediated vasoconstriction, thus monitoring the SPI during general anesthesia could lead to a reduced sympathetic response to surgical stimuli. Unfortunately there is not a desirable level of SPI, and it is unknown if difference in SPI values during the surgery might affect the postoperative outcome.

Intraoperative hemodynamic parameters and SPI will be recorded in conjunction with preoperative cardiovascular risk scores and will be used to develop a multiple variable model for postoperative risk of myocardial ischemic events.

In this study Electrocardiogram, invasive arterial pressure, photoplethysmography,and electroencephalographic entropy will be collected continuously from 10 min before induction of general anesthesia until 20 min after awakening from anesthesia. Gupta's score and Revised Cardiac Risk Index will be recorded the day before surgery.

Blood samples for high sensitive cardiac troponin T (hs-TnT) assay will be collected on day of surgery (baseline) and on postoperative day 1, 2 and 3. According to this methodology, in this study postoperative myocardial ischemic events will be defined as:

1. Myocardial Infarction according to the third universal definition (Thygesen K. et al. Third universal definition of myocardial infarction. Circulation 2012;126:2020-35 )
2. Myocardial Injury defined a hs-TnT plasmatic concentration of (i) 20-65 ng/L with an increase >5ng/L between baseline to days 1-3, or (ii) >65 ng/L, or (iii) a rise >50% between baseline and days 1-3 in case of renal insufficiency, all of them in absence of non-ischemic causes of troponin increase (sepsis, pulmonary embolism, electrical cardioversion and acute respiratory failure).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective non-cardiac vascular surgery under general anesthesia

Exclusion Criteria:

* Raynaud's phemomenon
* permanent atrial fibrillation or non sinus rhythm on ECG or ectopic beats >5% of normal sinus beats
* implanted with pacemaker
* any circulation problem in forefingers
* scheduled for postoperative ICU admission
* a new therapy with beta-blockers started <7 days before the surgery

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing general anesthesia for elective non-cardiac vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prediction of Postoperative Myocardial Ischemia | 72 hours after the surgery
  Cox's proportional model of preoperative cardiovascular risk scores and physiologic intraoperative variables for prediction of the occurrence of Postoperative Myocardial Ischemia

SECONDARY OUTCOMES:
prediction of postoperative myocardial ischemic events or stroke | 30 days
  Cox's proportional model of preoperative cardiovascular risk scores and physiologic intraoperative variables for prediction of postoperative myocardial ischemic events or stroke
mortality | 30 and 90 days
  measured by clinical record review and phone interview

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Fatebenefratelli Sacco, Luigi Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
de-identified patients' data will be available to other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: after the publication of the study results
Access Criteria: researchers that have been approved by the principal investigator and by Ethical Committee

REFERENCES:
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Background] Mackey WC, Fleisher LA, Haider S, Sheikh S, Cappelleri JC, Lee WC, Wang Q, Stephens JM. Perioperative myocardial ischemic injury in high-risk vascular surgery patients: incidence and clinical significance in a prospective clinical trial. J Vasc Surg. 2006 Mar;43(3):533-8. doi: 10.1016/j.jvs.2005.11.013. PMID 16520168
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] van Waes JA, Nathoe HM, de Graaff JC, Kemperman H, de Borst GJ, Peelen LM, van Klei WA; Cardiac Health After Surgery (CHASE) Investigators. Myocardial injury after noncardiac surgery and its association with short-term mortality. Circulation. 2013 Jun 11;127(23):2264-71. doi: 10.1161/CIRCULATIONAHA.113.002128. Epub 2013 May 10. PMID 23667270
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, Ford I, Gonzalez-Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luscher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Sousa-Uva M, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014 Sep 14;35(35):2383-431. doi: 10.1093/eurheartj/ehu282. Epub 2014 Aug 1. No abstract available. PMID 25086026
- [Background] Biccard BM, Rodseth RN. Utility of clinical risk predictors for preoperative cardiovascular risk prediction. Br J Anaesth. 2011 Aug;107(2):133-43. doi: 10.1093/bja/aer194. Epub 2011 Jun 30. PMID 21719480
- [Background] Bergmann I, Gohner A, Crozier TA, Hesjedal B, Wiese CH, Popov AF, Bauer M, Hinz JM. Surgical pleth index-guided remifentanil administration reduces remifentanil and propofol consumption and shortens recovery times in outpatient anaesthesia. Br J Anaesth. 2013 Apr;110(4):622-8. doi: 10.1093/bja/aes426. Epub 2012 Dec 5. PMID 23220856
- [Background] Bergmann I, Szabanowski T, Brauer A, Crozier TA, Bauer M, Hinz JM. Remifentanil added to sufentanil-sevoflurane anesthesia suppresses hemodynamic and metabolic stress responses to intense surgical stimuli more effectively than high-dose sufentanil-sevoflurane alone. BMC Anesthesiol. 2015 Jan 18;15(1):3. doi: 10.1186/1471-2253-15-3. eCollection 2015. PMID 25670917
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Colombo R, Marchi A, Borghi B, Fossali T, Tobaldini E, Guzzetti S, Raimondi F. Influence of gravitational sympathetic stimulation on the Surgical Plethysmographic Index. Physiol Res. 2015;64(2):183-9. doi: 10.33549/physiolres.932798. Epub 2014 Oct 15. PMID 25317683
- [Background] Colombo R, Marchi A, Borghi B, Fossali T, Rech R, Castelli A, Corona A, Guzzetti S, Raimondi F. Pulse Photoplethysmographic Analysis Estimates the Sympathetic Activity Directed to Heart and Vessels. Anesthesiology. 2015 Aug;123(2):336-45. doi: 10.1097/ALN.0000000000000712. PMID 26035252
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280